CLINICAL TRIAL: NCT00002971
Title: A Phase I Trial of Pre-Surgical O6-Benzylguanine in the Treatment of Patients With Malignant Glioma
Brief Title: O(6)-Benzylguanine in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NABTC-9702; CDR0000065479 (Registry Identifier: PDQ (Physician Data Query)); NCI-T96-0103
Record Dates: First submitted 1999-11-01; First posted 2003-05-05 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult anaplastic astrocytoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Astrocytoma; Gliosarcoma | interventions — O(6)-benzylguanine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: O6-benzylguanine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of O(6)-benzylguanine given before surgery to patients who have malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose of O6-benzylguanine (O6-BG) that produces total depletion of tumor O6-alkylguanine-DNA alkyltransferase (AGT) levels in more than 90% of patients with cerebral anaplastic astrocytoma or glioblastoma multiforme.
* Determine the qualitative and quantitative toxicities of O6-BG in this patient population.

OUTLINE: This is a dose escalation study.

Part I: The first cohort of 10 patients receives O6-benzylguanine (O6-BG) IV over 1 hour at dose level 1 beginning 6 hours prior to surgery. If at least 3 of 10 patients in the first cohort have detectable levels of O6-alkylguanine-DNA alkyltransferase (AGT), then a second cohort of 10 patients receives O6-BG as above at dose level 2. Dose escalation continues until at least 8 of 10 patients have undetectable AGT activity. At this point, 4 additional patients are accrued. If at least 11 of 14 patients at this dose level have undetectable levels of AGT, then this dose level constitutes the biologic modulatory dose of O6-BG. If less than 11 of 14 patients have undetectable levels of AGT, then 10 additional patients are treated at a higher dose. If at any time 3 or more patients at a dose level have detectable AGT activity, accrual is stopped at that dose level and patients are treated at the next higher dose level. (Part I closed to accrual effective 7/10/2000)

Part II: An additional cohort of 14 patients receives O6-BG at dose level 5 beginning 18 hours prior to surgery.

PROJECTED ACCRUAL: Part I of this study closed to accrual effective 7/10/2000. A total of 14 patients will be accrued for part II of this study at a rate of 3 patients per month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Must be undergoing a diagnostic/therapeutic craniotomy for biopsy/resection of recurrent or newly diagnosed (or presumed) cerebral anaplastic astrocytoma or glioblastoma multiforme

  * Patients undergoing stereotactic biopsy or partial resection are eligible

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* SWOG 0-2 OR
* Karnofsky 60-100%

Hematopoietic:

* WBC at least 3,500/mm3
* Absolute neutrophil count at least 1,800/mm3
* Platelet count at least 125,000/mm3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT less than 2 times upper limit of normal

Renal:

* Creatinine less than 1.5 mg/dL OR
* Creatinine clearance greater than 70 mL/min

Cardiovascular:

* No cardiovascular illnesses that cannot be adequately controlled with
* appropriate therapy or would increase risk, e.g.:
* Severe cardiac disease such as uncontrolled arrhythmias or conduction
* defects
* Major problems with edema (e.g., residual leg swelling from deep venous
* thrombosis)
* Recent coronary artery disease
* Poorly controlled hypertension (systolic pressure greater than 180 mm Hg,
* diastolic pressure greater than 110 mm Hg)

Other:

* No other medical illnesses that cannot be adequately controlled with
* appropriate therapy or would increase risk, e.g.:
* Major problems with edema (e.g., Cushing's syndrome)
* Major psychiatric illness
* No other malignancy requiring active therapy
* Not pregnant or nursing
* Fertile patients must us effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Must have failed or received no prior treatment with a nitrosourea,
* procarbazine, or temozolomide
* No prior O6-benzylguanine
* At least 4 weeks since prior chemotherapy and recovered

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 6 weeks since prior radiotherapy
* No prior radiotherapy to greater than 10-20% of bone marrow

Other:

* No concurrent therapy for any other malignancy
* At least 2 weeks since other prior investigational drug

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-06-19 (Actual); Primary Completion 2003-02-20 (Actual); Study Completion 2009-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Prados, MD, Study Chair — UCSF Medical Center at Parnassus
Locations (9):
- United States (9):
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin